CLINICAL TRIAL: NCT03365232
Title: Chairside Time and Bond Failure of Non Custom Versus Custom Base Orthodontic Attachments During Indirect Bonding: A Randomized Clinical Trial
Brief Title: Chairside Time and Bond Failure of Non Custom Versus Custom Base Orthodontic Attachments During Indirect Bonding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Saied Mahmoud Hassan, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CEBC-CU-2017-11-13
Record Dates: First submitted 2017-11-25; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non custom base attachment (Experimental)
  Interventions: Device: non custom base attachment
- custom base attachment (Active Comparator)
  Interventions: Device: custom base attachment

INTERVENTIONS:
Device: non custom base attachment — non custom base attachment
  Arms: non custom base attachment
Device: custom base attachment — custom base attachment
  Arms: custom base attachment

SUMMARY:
compare the chair side time, clinical orthodontic attachment bond failure and accuracy of transfer between non custom attachment base and custom attachment base indirect techniques.

ELIGIBILITY:
Inclusion Criteria:

- Patients should have

1. Maxillary sound teeth and undergoing fixed orthodontic treatment.
2. Space problems ranging from spacing to mild crowding.
3. Good oral hygiene.

Exclusion Criteria:

1. Patients with partially erupted teeth in the maxillary arch .
2. Signs of caries, large restorations fluorosis, hypoplasia or abnormalities of crown morphology.
3. The need of banding.
4. Bad oral hygiene measures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
chair side time | an average of 30 minutes
  using stopwatch

SECONDARY OUTCOMES:
immediate bond failure | immediately after bonding
  number of debonded attachments using hand instrument pressure

OTHER OUTCOMES:
accuracy of orthodontic attachments transfer | one day after bonding
  linear (mm) scale using geomagic software
accuracy of orthodontic attachments transfer | one day after bonding
  angular (degrees) scale using geomagic software